CLINICAL TRIAL: NCT04142697
Title: Visual and Vestibular Percepts of Motion
Brief Title: Human Visual and Vestibular Motion Perception Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Benjamin Crane, Associate Professor, University of Rochester
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 3911; R01DC013580 (NIH)
Record Dates: First submitted 2019-10-21; First posted 2019-10-29 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Vestibular Disease
MeSH Terms: conditions — Vestibular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy subjects (Active Comparator)
  Interventions: Behavioral: Heading direction adaptation
- Vestibular Disease patients (Active Comparator)
  Interventions: Behavioral: Heading direction adaptation

INTERVENTIONS:
Behavioral: Heading direction adaptation — Will adapt subject's perceived heading direction using exposure to visual environments that include rotation and situations where visual and inertial heading direction are systematically offset.

SUMMARY:
The purpose this study is to measure sensitivity to visual and vestibular or balance motion. It is hoped that the results may help researchers better understand how aging and disease affect motion perception.

DETAILED DESCRIPTION:
As people move through natural environments, they experience both visual and inertial stimuli. These can be integrated into a unified perception of self-motion (i.e. common causation) or segregated so that inertial or vestibular stimuli represents self-motion and visual represents external motion. There has been very little work on how causal inference (CI) or determination of common causation occurs for visual and inertial stimuli. Yet this is an important factor in fall risk, motion sickness, simulator sickness, concussion, dementia, and migraine. This proposal aims to develop and establish methods for studying CI in visual and inertial heading perception. This will be used to define the relevant variables in CI for these sensory systems. Common causation is likely a plastic process that occurs when stimuli occur simultaneously. The proposal will also examine this hypothesis by adapting heading perception, which may form the basis for a novel vestibular rehabilitation method.

Aim I: Causal inference (CI) for visual and inertial headings. During natural movements visual and inertial cues occur together. Inertial cues always represent self-motion, visual cues are ambiguous as they can represent motion through a fixed environment, environmental motion relative to the observer, or a combination of both. IA. Techniques for measuring CI for visual and inertial stimuli are not well established. The investigators have developed a technique to measure CI by presenting offset visual and inertial headings simultaneously using a full range of possible directions within the horizontal plane. Subjects report the perceived direction of the visual and inertial stimuli independently and whether or not they share common causation. These trial blocks can be repeated to determine reproducibility. IB. Parameters that influence perception of CI will be varied to determine their relative influences. These parameters will include stimulus timing, duration, and visual field size. It is hypothesized that full-field visual stimuli that are most consistent with the inertial stimulus will be perceived as having common causation. IC. Subjects with unilateral vestibular lesions will be tested using the techniques in IA. These individuals may have increased reliance on visual cues as well as decrease reliability and biases in inertial heading perception. As such, this may cause inertial headings to be more influenced by vision and result in a greater range of common causation.

Aim II: Visual-inertial heading adaptation. Plasticity in vestibular perception has received minimal attention, despite perception being the primary issue in common disorders such as vertigo, motion, and simulator sickness. Better understanding of how adaptation occurs could form the basis for improved therapeutic options as well as better tolerated virtual environments and simulations. IIA. Exposure to visual and inertial headings with similar characteristics, that are systematically offset, will be studied. It is hypothesized that exposure to this situation will influence subsequent visual and inertial heading perception as well as their common causation. These factors will also be measured before and after adaptation. The limits of what types of offsets can induce adaptation, and the range of headings that can be adapted will be explored. IIB. Preliminary data demonstrate that heading adaptation can also be induced by exposure to a virtual environment with an angular velocity offset in the visual stimulus. This method of adaptation will also be studied with regard to its influence on perception of rotation, visual and inertial headings and common causation of these headings. As with IIA, the potential limitations of the method will be explored.

Aim III: Heading adaptation after vestibular loss. Errors in heading perception are a clinically significant problem. Abnormal perception of rotation often quickly normalizes after vestibular lesions, but preliminary data indicate heading perception remains deviated for years afterwards. This could be due to asymmetry in the otolith system which current vestibular rehabilitation methods do not address. Abnormal heading perception may be a significant factor in other disorders including vestibular migraine, dementia, and concussion. Understanding long-term adaptation is potentially important in these populations. IIIA. Time course and etiology of perceptual pathology after acute vestibular lesions is unclear. This will be investigated by sequentially measuring bias and perceptual thresholds of yaw rotation, sway, and heading in individuals with acute loss of vestibular function. Initially subjects have a rotation bias towards the intact side which normalizes over time. The heading bias may correlate with rotational bias or may be related to otolith dysfunction, as measured with sway translation perception, or may occur as a result of adapting to the rotatory vertigo. IIIB. Study of long-term heading adaptation in subjects with chronic unilateral vestibular hypofunction (e.g. those who have had vestibular schwannomas removed, gentamicin ablative therapy for Meniere's disease). Since these subjects often have biased heading perception at baseline, they may be able to exhibit long term adaptation. Heading perception as well as visual-inertial common causation will be measured using the techniques described in Aim IC. Ability to adapt these patients to heading offsets will be measured using the methods established in normal controls (Aim II) but the adaptation will always be in a consistent direction to attempt to normalize baseline deviation in heading perception. It will be determined if durable long-term heading adaptation can be achieved. The proposal aims to understand how visual and inertial cues inform motion perception and how adaptation has the potential to improve pathological perception.

ELIGIBILITY:
Inclusion Criteria:

Healthy subjects:

* general good health

Vestibular Disease patients:

* general good health
* specific unilateral or bilateral vestibular loss

Exclusion Criteria:

Healthy subjects:

* subjects who are institutionalized or otherwise not self-sufficient.
* enduring sequelae due to diseases of the nervous system, eyes, ears, head and neck, and limbs, except for changes commensurate with normal aging (e.g. presbyacusic hearing loss, mild cataract, etc.).
* abnormal cognitive function, which if in question can be determined as a score of <27 on the Mini-Mental State test.
* corrected visual acuity worse than 20/20 up to age 65, worse than 20/40 if >65
* abnormal binocular stereo-acuity or visual fields.
* any defects in cranial nerve, oculomotor, cerebellar/coordination, and somatosensory functions.
* any abnormal oculomotor and vestibular function (caloric tests)

Vestibular Disease patients:

* Inability to perform the study tasks due to sensory, motor, or postural limitations

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-09-15 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Mean Heading perception | Baseline to 1 week
  Heading perception will be measured using two alternative forced choice and magnitude estimation procedures and reported in degrees. It is measured in degrees of azimuth with positive to the right and negative to the left of straight ahead (defined as 0 degrees).

SECONDARY OUTCOMES:
Change in Mean Dizziness Handicap Inventory (DHI) | Baseline to 1 week
  The (DHI) will be measured in subjects with unilateral vestibular hypo function to ensure symptoms are not worsening, but will not be measured in health subjects. This is a a 25 question scale ranging from 0-100 with 100 indicating worse dizziness.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data provided upon request to principal investigator